CLINICAL TRIAL: NCT04940390
Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of STS101 (Dihydroergotamine Nasal Powder) in the Acute Treatment of Migraine
Brief Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Assess STS101 in the Acute Treatment of Migraine
Acronym: SUMMIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Satsuma Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STS101-007
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura
Keywords: dihydroergotamine; dihydroergotamine mesylate; migraine
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura | interventions — Dihydroergotamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- STS101 (Experimental): STS101 (dihydroergotamine nasal powder)
  Interventions: Drug: Dihydroergotamine
- STS101 Placebo (Experimental): STS101 Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dihydroergotamine — Dihydroergotamine is a semi-synthetic derivative of ergotamine tartrate.
  Other Names: Dihydroergotamine Mesylate
  Arms: STS101
Drug: Placebo — Placebo for STS101
  Other Names: STS101 Placebo
  Arms: STS101 Placebo

SUMMARY:
Study STS101-007 is a randomized, double-blind, parallel group, placebo-controlled, multicenter study to evaluate the efficacy, safety, and tolerability of single doses of STS101 (dihydroergotamine nasal powder) in the acute treatment of migraine.

DETAILED DESCRIPTION:
Study STS101-007 is a multi-center, single-dose, randomized, double-blind, placebo-controlled, parallel group study in subjects with acute migraine (ages 18 to 65 years).

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females, 18-65 years of age at the time of Screening Visit
* Subject has at least 1-year history of migraines (with or without aura), according to the International Classification of Headache Disorder, 3rd Edition (ICHD3)

Key Exclusion Criteria:

* Pregnant or breast-feeding women
* Women of child-bearing potential not using or not willing to use highly effective contraception.
* Diagnosis of headache conditions other than migraine with or without aura, including diagnosis of basilar or hemiplegic migraines or cluster headache.
* History of coronary artery disease, coronary artery vasospasm (including Printz-metals' angina), clinically significant arrhythmia or, peripheral vascular disease, ischemic disease (e.g. Raynaud's syndrome, ischemic bowel syndrome, angina pectoris, myocardial infarction, or documented silent ischemia); percutaneous coronary intervention, or cardiac surgery.
* History of cerebrovascular disease, including but not limited to stroke, transient ischemic attack, cerebral hemorrhage, subarachnoid hemorrhage.
* Diagnosis of major depression with current symptoms, psychosis, alcohol abuse or dependence, drug abuse or dependence, major psychiatric conditions (e.g. schizophrenia, psychosis or Bipolar disorder), dementia. Other significant neurological or psychiatric disorders (including other pain syndromes or risk of suicide) that in the opinion of the investigator might interfere with study participation and assessments or subject safety.
* Any clinically significant symptoms or conditions, including but not limited to central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator might interfere with study assessments or safety of participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1591 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Albrecht, MD, Study Chair — Satsuma Pharmaceuticals, Inc.
Locations (127):
- United States (127):
  - MD First Research, Chandler, Arizona
  - Elite Clinical Studies, Phoenix, Arizona
  - Alliance For Multispecialty Research, Tempe, Arizona
  - Cognitive Clinical Trials, LLC, Tempe, Arizona
  - Clinedge, LLC, Tucson, Arizona
  - ERG Clinical, Little Rock, Arkansas
  - Hope Clinical Research, Canoga Park, California
  - Wr-Pri, Llc, Encino, California
  - Neuro-Pain Medical Center Ince, Fresno, California
  - Estudy Site - La Mesa, La Mesa, California
  - Wr-Pri Llc, Los Alamitos, California
  - Downtown LA Research Center, Los Angeles, California
  - Clinical Research Institute, Los Angeles, California
  - Wr-Pri Llc, Newport Beach, California
  - Artemis Institute for Clinical Research - San Diego, San Diego, California
  - WR-MCCR, San Diego, California
  - Acclaim Clinical Research, San Diego, California
  - National Research Institute, A Clinical Research Organization, Santa Ana, California
  - Alpine Clinical Research Center, Inc, Boulder, Colorado
  - Clinedge, LLC, Cromwell, Connecticut
  - Neurology Offices of South Florida, Boca Raton, Florida
  - Velocity Clinical Research, Hallendale Beach, Hallandale, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Elite Research Network, LLC a Florida LLC, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Elite Research Network LLC a Florida LLC, Jupiter, Florida
  - Multi-Specialty Research Associates, Lake City, Florida
  - Clinicloud, Maitland, Florida
  - Next Phase Research, Miami, Florida
  - Applemed Research Group, Miami, Florida
  - Biotech Pharmaceuticals Group LLC, Miami, Florida
  - Novel Clinical Research Center LLC, Miami, Florida
  - Floridian Research, Miami, Florida
  - Behavioral Clinical Research, North Miami, Florida
  - Accel-Orange City, Orange City, Florida
  - CNS Health Care Orlando, Orlando, Florida
  - Complete Health Research, Ormond Beach, Florida
  - Oveido Medical Research, Oviedo, Florida
  - Santos Research Center, Tampa, Florida
  - VICIS Clinical Research, Inc, Tampa, Florida
  - Palm Beach Research, West Palm Beach, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - Delricht, Atlanta, Georgia
  - I-Research Atlanta, Decatur, Georgia
  - Alpha Clinical Research Georgia, Johns Creek, Georgia
  - Clin-Edge, LLC, Marietta, Georgia
  - I Research Savannah, Savannah, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - CIS Research, Wauconda, Illinois
  - Medisphere Medical Research Center, Evansville, Indiana
  - PMG Research Inc, Ames, Iowa
  - Meridian Clinical Research, Sioux City, Iowa
  - Integrated Clinical Trial SVC, West Des Moines, Iowa
  - Alliance For Multispecialty Research, Lexington, Kentucky
  - Louisville Metabolic & Atherosclerosis Research Center, Louisville, Kentucky
  - Delricht Research, Baton Rouge, Louisiana
  - Crescent City Headache and Neurology, Chalmette, Louisiana
  - Delricht, Covington, Louisiana
  - Alliance for Multispecialty Research, New Orleans, Louisiana
  - Delricht-New Orleans, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - BTC of New Bedford, New Bedford, Massachusetts
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - "Medvadis Research Corp, Llc @Boston Paincare Center ", Waltham, Massachusetts
  - MHNI, Ann Arbor, Michigan
  - Minneapolis Clinic of Neurology, Burnsville, Minnesota
  - Delricht, Gulfport, Mississippi
  - Alliance for Multispecialty Research, Kansas City, Missouri
  - Montana Medical Research, Inc, Missoula, Montana
  - Skyline Medical Center, PC CCT Research, Elkhorn, Nebraska
  - Cognitive Clinical Trials, LLC, Fremont, Nebraska
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Wake Research-Clinical Research Center of Nevada LLC, Las Vegas, Nevada
  - Clinedge LLC, North Las Vegas, Nevada
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Integrative Clinical Trials, Brooklyn, New York
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - North Suffolk Neurology, Commack, New York
  - Drug Trials America, Hartsdale, New York
  - Central New York Clinical Research, Manlius, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - PMG Research of Charlotte, Charlotte, North Carolina
  - Onsite Clinical, Charlotte, North Carolina
  - Headache Wellness Center - Greensboro, Greensboro, North Carolina
  - Pharmquest, LLC, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - PMG Research, Inc, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research Inc, Winston-Salem, North Carolina
  - Plains Clinical Research, South West Fargo, North Dakota
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Aventiv Research, Columbus, Ohio
  - Aventiv Research, Inc, Dublin, Ohio
  - OK Clinical Research, Edmond, Oklahoma
  - Elite Research Network, LLC a Florida LLC, Norman, Oklahoma
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Delricht Research, Tulsa, Oklahoma
  - Tekton Research, Yukon, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Ocean State Clinical Research Partners, Lincoln, Rhode Island
  - Velocity Clinical Research.- Providence, Warwick, Rhode Island
  - Clinedge LLC - Clinical Trials SSC, Charleston, South Carolina
  - Tribe CR, Greenville, South Carolina
  - Coastal Carolina Research Center Inc, North Charleston, South Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - Future Search Trials of Neurology, Austin, Texas
  - Premier Family Physicians, Austin, Texas
  - Discoveresearch, Bryan, Texas
  - Future Search Trials of Dallas, LP, Dallas, Texas
  - Cedar Health Research, LLC, Dallas, Texas
  - North Texas Institute of Neurology, Frisco, Texas
  - Epic Clinical Research, Lewisville, Texas
  - DM Clinical Research, Magnolia, Texas
  - Village Health Partners, Plano, Texas
  - Sun Research, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Advanced Research Institute, Ogden, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Alliance For Multispecialty Research, Norfolk, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Womens, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1591 participants were randomized in the study, of which 1424 reported a qualifying migraine attack, received study drug, and reported efficacy data in at least one post-treatment e-diary (modified intent to treat population).
Groups:
- STS101 5.2 mg: Subjects received a single oral dose of STS101 (dihydroergotamine nasal powder) 5.2 mg
- STS101 Placebo: Subjects received a single oral dose of Placebo for STS101 (dihydroergotamine nasal powder)
Period: Overall Study
Arm/Group | STS101 5.2 mg | STS101 Placebo
Started | 796 | 795
Modified Intent-to Treat Population | 716 | 708
Safety Population | 731 | 729
Completed | 771 | 770
Not Completed | 25 | 25

BASELINE CHARACTERISTICS:
Population: Patient demographics are presented for the mITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | STS101 5.2 mg | STS101 Placebo | Total
Number analyzed (Participants) | 716 | 708 | 1424
Age, Customized [Count of Participants; unit: Participants]
  18-35 years | 312 | 297 | 609
  >35-50 years | 286 | 283 | 569
  >50-65 years | 118 | 128 | 246
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 567 | 564 | 1131
  Male | 149 | 144 | 293
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 8
  Asian | 25 | 24 | 49
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 86 | 97 | 183
  White | 591 | 576 | 1167
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 716 | 708 | 1424

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Freedom From Migraine Headache Pain at 2 Hours Post Dose
Description: The subject's rating was documented on a four-point scale from no pain (= 0), mild pain (= 1), moderate pain (= 2) to severe pain (= 3). Pain freedom means the pain went from moderate (2) or severe (3) to no pain (0).
Time Frame: 2 Hours Post-Dose
Population: The analysis was performed on the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | STS101 5.2 mg | STS101 Placebo
Number analyzed (Participants) | 716 | 708
Participants | 146 | 124

2. Primary Outcome: Percentage of Subjects With Freedom From Most-Bothersome Symptom at 2 Hours Post Dose
Description: Subjects were prompted to document the presence of 3 symptoms (photophobia, phonophobia, and nausea) immediately before study drug administration and during the treated migraine attack.
Time Frame: 2 Hours Post-Dose
Population: This analysis was conducted on the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | STS101 5.2 mg | STS101 Placebo
Number analyzed (Participants) | 716 | 708
Participants | 265 | 230

3. Secondary Outcome: Percentage of Subjects With Relief From Migraine Headache Pain at 2 Hours Post Dose
Description: The subject's rating was documented on a four-point scale from no pain (= 0), mild pain (= 1), moderate pain (= 2) to severe pain (= 3). Pain relief means the pain went from moderate (2) or severe (3) to mild pain (1) or no pain (0).
Time Frame: 2 Hours Post Dose
Population: This analysis was conducted on the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | STS101 5.2 mg | STS101 Placebo
Number analyzed (Participants) | 716 | 708
Participants | 379 | 316

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the date of randomization up to the end of subject's participation in the study which was no later than Study Day 66. Serious adverse events (SAEs) were collected from the date of informed consent up to the end of subject's participation in the study which was no later than Study Day 66.
Description: The safety population was used for adverse event reporting.
Arm/Group | STS101 5.2 mg | STS101 Placebo
All-Cause Mortality (participants affected / at risk) | 0/731 | 0/729
Serious Adverse Events (participants affected / at risk) | 3/731 | 0/729
Other Adverse Events (participants affected / at risk) | 111/731 | 14/729
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STS101 5.2 mg (N=731) | STS101 Placebo (N=729)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Procedural Abdominal Pain Post-hysterectomy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asthma Exacerbation/Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | STS101 5.2 mg (N=731) | STS101 Placebo (N=729)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 61 | 11
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 23 | 1
Dysgeusia (Nervous system disorders) | 27 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT04940390/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT04940390/SAP_001.pdf